CLINICAL TRIAL: NCT03466203
Title: A 12 Week Phase Ib Randomized Investigator and Subject Blinded Placebo Controlled Repeat-dose Study of LLF580
Brief Title: Safety Study of LLF580 in Obese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLLF580X2102
Record Dates: First submitted 2018-02-09; First posted 2018-03-15 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: obesity; hypertriglyceridemia
MeSH Terms: conditions — Obesity; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LLF580 (Experimental): LLF580 every 28 days * 3
  Interventions: Biological: LLF580
- Placebo (Placebo Comparator): Placebo to LLF580 every 28 days * 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: LLF580 — LLF580 300mg
  Arms: LLF580
Drug: Placebo — Placebo to LLF580
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple doses of LLF580 administered subcutaneously over 3 months in obese subjects. In addition, the study will also determine early efficacy signals in various metabolic diseases associated with elevated triglycerides and/or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range of 30 to 45 kg/m2, inclusive, with ethnic adjustment (≥27.5 kg/m2 for Asian individuals).
* Fasting triglyceride 150 - 500 mg/dL (1.69 - 5.65 mmol/L), inclusive, at screening.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* History of hepatobilliary disease.
* Liver disease or liver injury as indicated by abnormal liver function tests.
* Chronic infection with Human Immunodeficiency Virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV).
* Fasting triglycerides greater than or equal to 500 mg/dL [5.65 mmol/L], or concomitant use of drug treatment for hypertriglyceridemia (fibrates, omega-3 fatty acids, nicotinic acid).
* History of pancreatic injury or pancreatitis.
* History of hypersensitivity to drugs of similar biological class, FGF21 protein analogue, or Fc fusion proteins.
* History of bone disorders or low vitamin D level.
* Contraindications to MRI.
* Change in body weight (more than 5% self-reported OR 5 kg self-reported change during the previous 3 months).
* Use of weight loss drugs.
* Enrollment in a diet, weight loss or exercise programs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability following repeated dosing of LLF580 | 12 weeks
  To assess the safety and tolerability in obese subjects following repeated dosing of LLF580 by subcutaneous (SC) injection over 12 weeks.

SECONDARY OUTCOMES:
LDL-C, HDL-C | 12 weeks
  To assess the effects of LLF580 on lipid profiles.
serum CTX-1, P1NP, and osteocalcin | 12 weeks
  To assess the potential effects of LLF580 on these biomarkers.
Body weight | 12 weeks
  To assess the effects of LLF580 on weight.
BMI | 12 weeks
  To assess the effects of LLF580 on BMI
serum BSAP | 12 weeks
  To assess the potential effects of LLF580 on these biomarkers.
urine NTX-1 | 12 weeks
  To assess the potential effects of LLF580 on these biomarkers.
Total cholesterol | 12 weeks
  To asses the effects of LLF580 on lipid profiles
Triglycerides (fasting) | 12 weeks
  To assess the effects of LLF580 on lipid profiles

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rader DJ, Maratos-Flier E, Nguyen A, Hom D, Ferriere M, Li Y, Kompa J, Martic M, Hinder M, Basson CT, Yowe D, Diener J, Goldfine AB; CLLF580X2102 Study Team. LLF580, an FGF21 Analog, Reduces Triglycerides and Hepatic Fat in Obese Adults With Modest Hypertriglyceridemia. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e57-e70. doi: 10.1210/clinem/dgab624. PMID 34431493
- See also: Results for CLLF580X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17731
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=649